CLINICAL TRIAL: NCT05286957
Title: Minimal Residual Disease (MRD)-Guided Adjuvant Tislelizumab and Chemotherapy in Resected Stage IIA-IIIB Non-small Cell Lung Cancer (NSCLC): a Randomized Controlled Phase II Study (Seagull)
Brief Title: MRD-guided Adjuvant Tislelizumab and Chemotherapy in Resected Stage IIA-IIIB NSCLC
Acronym: Seagull
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Collaborators: BeiGene (Industry)
Responsible Party: Principal Investigator, Qi Yu, chief physician, The First Affiliated Hospital of Zhengzhou University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L2021-Y471
Record Dates: First submitted 2022-03-01; First posted 2022-03-18 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: NSCLC
Keywords: ctDNA-MRD
MeSH Terms: interventions — Drug Therapy; Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MRD-guided adjuvant tislelizumab and chemotherapy (Experimental): MRD+: Tislelizumab 200mg Q3W + chemotherapy 1-4 cycles and followed by Tislelizumab 200mg Q3W Up to 16 cycles or until PD or intolerable toxicity or withdrawal
  MRD-: Adjuvant chemotherapy and surveillance the MRD status, the patient will receive treatment for MRD+ patient when MRD detected,
  Interventions: Drug: adjuvant tislelizumab and chemotherapy for MRD+ patients
- Non MRD-guided adjuvant tislelizumab and chemotherapy (Active Comparator): patients in non MRD-guided arm receive adjuvant tislelizumab and chemotherapy
  Interventions: Drug: adjuvant tislelizumab and chemotherapy for MRD+ patients; Drug: adjuvant chemotherapy for MRD- patients

INTERVENTIONS:
Drug: adjuvant tislelizumab and chemotherapy for MRD+ patients — MRD+ patients receive adjuvant tislelizumab and chemotherapy while MRD- patients just is recommended receive adjuvant chemotherapy untill be detected MRD+
  adjuvant tislelizumab and chemotherapy (cisplatin/carboplatin + paclitaxel or cisplatin/carboplatin + pemetrexed,dependent on tumor histology and at investigator's discretion)
Drug: adjuvant tislelizumab and chemotherapy for MRD+ patients — patients receive adjuvant tislelizumab and chemotherapy regardless of MRD status
  Arms: MRD-guided adjuvant tislelizumab and chemotherapy
Drug: adjuvant chemotherapy for MRD- patients — MRD- patients just be recommended receive adjuvant chemotherapy untill be detected cisplatin/carboplatin + paclitaxel or cisplatin/carboplatin + pemetrexed,dependent on tumor histology and at investigator's discretion, limited to ≤4 cycles
  Arms: Non MRD-guided adjuvant tislelizumab and chemotherapy

SUMMARY:
Seagull is a phase Ⅱ study designed to investigate the efficacy and safety of MRD-guided adjuvant tislelizumab and chemotherapy vs adjuvant tislelizumab and chemotherapy in patients with resectable NSCLC

DETAILED DESCRIPTION:
In the phase II trial, the efficacy and safety of MRD-guided adjuvant tislelizumab and chemotherapy will be compared with that of standard adjuvant tislelizumab and chemotherapy in patients with resectable NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with age ≥ 18 years old, gender is not limited.
2. Histologically confirmed primary NSCLC, postoperative stage is IIA, IIB, IIIA or T3N2IIIB.
3. Receiving complete resection
4. Paraffin-embedded sections (10-15 pieces) or fresh frozen tissue are required.
5. ECOG score of 0 or 1.
6. Females of childbearing age should take appropriate contraceptive measures from screening to 3 months after discontinuation of study treatment and should not breastfeed. The pregnancy test was negative before starting dosing.
7. Male patients should use barrier contraception from screening to 3 months after discontinuation of study treatment.
8. The subjects themselves participated voluntarily and signed the informed consent in writing.

Exclusion Criteria:

1. The patient has received immune checkpoint inhibitors such as anti-PD-1, PD-L1 or CTLA-4, other immunotherapy or systemic immune modulators (including but not limited to interferon, IL-2 and TNF etc).
2. Histopathology with small cell or large cell endocrine tumor component.
3. Harboring EGFR sensitizing mutation or ALK gene translocation
4. History of other malignant tumors, except for non-melanoma skin cancer, carcinoma in situ or other solid tumors that have been effectively treated, and no evidence of any disease for >5 years after the last treatment.
5. At the start of the study treatment, there are residual toxicities of the previous treatment that are greater than CTCAE 1 and have not been alleviated, except for alopecia and grade 2 neurotoxicity caused by previous chemotherapy.
6. Any serious or uncontrolled systemic disease, including uncontrolled high blood pressure, active bleeding, active infection including hepatitis B, C, HIV, etc., which the investigator considers unsuitable to participate in the study or affect the trial program compliance.
7. History of ILD, drug-induced interstitial lung disease, radiation pneumonitis requiring steroid therapy, or any evidence of clinically active interstitial lung disease
8. Insufficient bone marrow reserve or organ function.
9. History of hypersensitivity reactions to any active or inactive ingredient of tislelizumab or to drugs that are chemically similar to tislelizumab or in the same class of tislelizumab.
10. Patients who, in the judgment of the investigator, may not comply with the procedures and requirements of the study.
11. Patients who, in the investigator's judgment, have any condition that compromises patient safety or interferes with the evaluation of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-20 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
2-year PFS rate | up to 36 months after enrollment or study close
  Progression-free survival (per RECIST 1.1) is defined as the time from the starting date of study drug to the date of first documentation of disease progression or death, whichever occurs first. Subjects who do not have disease progression will be censored at their last valid tumor assessment. PFS rate at 1 year as estimated by Kaplan-Meier method.

SECONDARY OUTCOMES:
Percentage of patients changed from MRD+ to MRD- after treatment with tislelizumab for 6 months，12 months | At the end of Cycle 8(each cycle is 21 days)、Cycle 16 (each cycle is 21 days)
  Percentage of patients changed from MRD+ to MRD- after treatment with Tislelizumab for 9 months，12months

CONTACTS AND LOCATIONS:
Overall Officials: Yu Qi, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- The First Affiliated Hospital of Zhengzhou University,, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided